CLINICAL TRIAL: NCT00512980
Title: A Randomized Phase II Study of Prednisone, Vinblastine, Doxorubicin, and Gemcitabine in Patients With Intermediate Stage Hodgkin's Lymphoma
Brief Title: PVAG-14 Pilot for Intermediate Stages Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lower recruitment rates as expected
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PVAG-14 pilot
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hodgkin Lymphoma
Keywords: intermediate stages
MeSH Terms: conditions — Hodgkin Disease | interventions — Prednisone; Vinblastine; Doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: prednisone; Drug: vinblastine; Drug: doxorubicin; Drug: gemcitabine
- 2 (Active Comparator)
  Interventions: Drug: prednisone; Drug: vinblastine; Drug: doxorubicin; Drug: gemcitabine

INTERVENTIONS:
Drug: prednisone
Drug: vinblastine
Drug: doxorubicin
Drug: gemcitabine

SUMMARY:
A randomized phase II study of prednisone, vinblastine, doxorubicin, and gemcitabine in patients with intermediate stage Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of Hodgkin's lymphoma
2. Stage

   * Clinical Stage IA, IB, IIA with at least one of the risk factors a-d given below
   * Clinical Stage IIB with one or both risk factors c-d given below risk factors:

     * Large mediastinal mass (≥ 1/3 of the greatest thorax diameter as measured by chest x-ray)
     * Extranodal involvement
     * High erythrocyte sedimentation rate (≥ 50 mm/h in patients without B-symptoms, ≥ 30 mm/h in patients with B-symptoms)
     * Three or more involved lymph node areas
3. No prior therapy for Hodgkin's lymphoma (exception: pre-phase treatment with corticosteroids and vinca-alkaloids for a maximum of seven days may not preclude trial participation if clinically indicated and all staging examinations have been performed; all forms of prior radiotherapy preclude trial participation)
4. Age: 18-60 years
5. Signed informed consent with understanding of the study procedures and the investigational nature of the study
6. Patient agrees that personal data and tissue samples are provided to the GHSG (protection of privacy as defined by law will be ensured)
7. Life expectancy > 3 months according to investigator judgement.

Exclusion Criteria:

1. Incomplete diagnosis of stage of disease
2. Prior or concurrent disease which prevents treatment according to protocol In particular the following contraindications:

   * Chronic obstructive pulmonary disease with global insufficiency
   * Symptomatic coronary heart disease
   * Cardiomyopathy or cardiac insufficiency (NYHA value of EF < 50% or FS < 25%)
   * Serious uncontrolled hypertension
   * Uncontrollable infection
   * Leucocyte concentration < 3.000/mm3 or thrombocyte concentration < 100.000/mm3
   * Creatinin clearance < 60 ml/min
   * Bilirubin > 2 mg/dl or GPT > 100 U/l or GOT > 100 U/I (exception: elevated values of Hodgkin's disease liver involvement)
   * HIV-Infection according to HIV test
   * Chronic or acute Hepatitis
3. HD as composite lymphoma
4. Prior chemotherapy or radiation
5. Malignant disease within the last 5 years (exceptions: basalioma, carcinoma in situ of the cervix uteri, completely resected melanoma TNMpT1)
6. Pregnancy, lactation, positive pregnancy test
7. Refusal to use effective contraception
8. WHO performance index > 2
9. Long-term ingestion of corticosteroids (e.g. for chronic polyarthritis) or antineoplastic drugs (e.g. methotrexate)
10. Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the trial and to formulate his/her own wishes correspondingly
11. Non compliance: Refusal of blood products during treatment, epilepsy, drug dependency, change of residence abroad, prior cerebral injury or similar circumstances which appear to make protocol treatment or long-term follow-up impossible
12. Antiepileptic treatment
13. General intolerance of any protocol medication
14. Any contraindication for study medication according to the summaries of product information
15. Simultaneous participation in another clinical
16. Institutionalization by law
17. Relation of dependence with the sponsor's representative / trialist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2008-08; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany